CLINICAL TRIAL: NCT05606211
Title: Pain in PASC - the Role of Sleep Disturbances
Brief Title: Pain in Long COVID-19: the Role of Sleep
Status: Active, not recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Monika Haack, Associate Professor of Neurology, Beth Israel Deaconess Medical Center
Other Study IDs: 2022P-000257
Record Dates: First submitted 2022-11-02; First posted 2022-11-04 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Long COVID: Individuals who have been infected with the corona virus and developed Long COVID
  Interventions: Other: No intervention
- No Long COVID: Individuals who have been infected with the corona virus and fully recovered.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational, no intervention

SUMMARY:
Pain is among the most frequently reported symptoms in Long COVID, along with sleep disturbances, fatigue, and cognitive impairments. Sleep plays a critical role in maintaining a pain-free state. The goal of this study is to characterize the type and severity of pain in Long COVID, to characterize sleep and sleep disturbances in Long COVID, and to understand the role of sleep in the development and persistence of pain symptoms in Long COVID.

ELIGIBILITY:
Inclusion Criteria:

* Females and males >18 years
* Confirmed history of SARS-CoV-2 infection

Exclusion Criteria

* History of chronic pain prior to SARS-CoV-2 infection
* Raynaud syndrome
* Pregnant/nursing

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have been infected with the corona virus and developed or did not developed Long COVID.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain reporting | 14 days
  Daily pain severity reporting on rating scale from 0 to 10 (greater values indicate greater pain)
Pain sensitivity | 1 day
  Pain thresholds to mechanical and temperature stimuli measured in kPa (pressure) and Celsius (heat). Lower values indicate lower pain thresholds.
Central pain modulation | 1 day
  Capacity of the CNS to modulate pain
Wearable based sleep characteristics | 2 weeks
  Estimation of sleep duration, fragmentation, regularity based on actigraphy
PSG based sleep characteristics | 1 day
  Sleep stages and architecture based on PSG

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Engert LC, Dang R, Daniel S, Bertisch SM, Maley JH, Fong TG, Serhan CN, Mullington JM, Haack M. Sleep disturbance affects inflammatory resolution in Long COVID. Prostaglandins Leukot Essent Fatty Acids. 2026 Feb 2;208:102728. doi: 10.1016/j.plefa.2026.102728. Online ahead of print. PMID 41650882